CLINICAL TRIAL: NCT05559801
Title: A Phase 1/2 Study to Examine the Safety and Preliminary Efficacy of Mesenchymal Stromal Cells on Linear Growth and Bone Health Parameters in Children With Type 3 Osteogenesis Imperfecta (OI)
Brief Title: Mesenchymal Cell Therapy in Osteogenesis Imperfecta (OI)
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Doris Fadoju, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003434
Record Dates: First submitted 2022-09-08; First posted 2022-09-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Osteogenesis Imperfecta; Osteogenesis Imperfecta Type III
MeSH Terms: conditions — Osteogenesis Imperfecta; Osteogenesis imperfecta, type 3

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Children with OI receiving Bone marrow-derived MSCs infusion (Experimental): Intravenously-infused allogeneic, bone marrow-derived mesenchymal stromal cells (MSCs) in children with Osteogenesis Imperfecta Type III that will be infused at 0 months, 4 months, 8 months, 12 months, 16 months, and 20 months, after enrollment.
  Interventions: Drug: Bone marrow-derived mesenchymal stromal cells (MSCs)

INTERVENTIONS:
Drug: Bone marrow-derived mesenchymal stromal cells (MSCs) — Mesenchymal stromal cells (MSCs) are cells of non-hematopoietic stromal origin that reside in bone marrow and a variety of tissues. MSCs will be prepared in a GMP Cell Production facility and administered to children age 3-10 years (at time of enrollment) with Osteogenesis Imperfecta Type III.
  Other Names: MSC infusions

SUMMARY:
This is a Phase 1/2 study to determine the safety and efficacy of allogeneic (third party), bone-marrow derived mesenchymal stromal cells (MSCs) for the treatment of Osteogenesis Imperfecta (OI) Type 3. It will evaluate this by looking at whether there are treatment related infusion reactions, and assessing linear growth rates and bone health, both of which are impaired in patients ages 3-10 with Osteogenesis Imperfecta Type 3. This is a single-site non-randomized clinical trial, that will take place at Children's Healthcare of Atlanta (CHOA) at Egleston and Emory Children's Center.

DETAILED DESCRIPTION:
This is a Phase 1/2 study to determine the safety and efficacy of allogeneic (third party), bone-marrow derived mesenchymal stromal cells (MSCs) for the treatment of Osteogenesis Imperfecta (OI) Type 3. It will evaluate this by looking at whether there are treatment related infusion reactions, and assessing linear growth rates and bone health, both of which are impaired in patients ages 3-10 with Osteogenesis Imperfecta Type 3. This is a single-site non-randomized clinical trial, that will take place at Children's Healthcare of Atlanta (CHOA) at Egleston and Emory Children's Center.

MSCs will be infused through IV every 4 months for 6 total infusions. There will be a baseline visit before MSC therapy is initiated, and there will be a follow up visits every 4 months for 1 year after the final MSC infusion. These infusions will take place in between pamidronate infusions (i.e. 2 months after the last pamidronate infusion, and 2 months before the next one). Pamidronate aids in treatment of bone pain and bone mineral density but does not correct the underlying defect nor does it show substantial improvements in linear growth.

After the MSC infusions, patients will be provided an overnight at Ronald McDonald House, or a hospital affiliated hotel so they can be near to the hospital in case of any unanticipated effects, and for a follow up visit the next morning.

Labs will be collected during every visit to look at bone metabolism. Limb and bone age x-rays, pQCT scans, and dual-energy x-ray absorptiometry (DXA) scans will be completed annually, while spine films will be completed every 18 months. These images will directly examine bone health. Body measurements will be taken every visit as well to assess linear growth. The patients' parents will complete events diaries and submit them each infusion day to evaluate fractures that occurred between visits. Patients and their parents will also complete quality of life surveys once a year.

There will be financial compensation for each study visit. Subjects will also be provided a free lunch on days when radiology visits occur and will be reimbursed for parking.

Subjects will be identified and recruited mainly through Children's endocrinology clinic. There will also be advertisements to the OI foundation, and neighboring pediatric hospitals with OI programs such as University of Alabama at Birmingham, and Vanderbilt. If identified as eligible to participate, the study team will seek approval by the subjects' primary endocrinologist. The consent process will then take place in person during a baseline visit.

There is an optional part of the study that involves donation of a bone fragment that is taken out during a routine surgical rodding procedure. This piece of bone is removed and discarded, if it is not donated, making it minimal risk. Bone sample donation will be available to OI Type 3 subjects receiving MSCs, and to OI Type 3 subjects who are not receiving MSCs but want to participate in research.

Leftover blood samples, and bone fragments may be stored for future research by the sponsor of this study.

The purpose of this study is to help doctors and scientists learn if serial MSC infusions will safely and effectively aid in growth, bone health, and ultimately improve motoric function and quality of life in this population.

ELIGIBILITY:
Inclusion Criteria:

* 1. Parent/legal guardian must be willing to sign consent forms to participate in this trial 2. Participants must be >3 years of age and <10 years of age at time of enrollment 3. Must carry mutation in either COL1A1 or COL1A2 genes and based on clinical assessment have severe Type 3 OI* 4. Must be pre-pubertal to minimize potential influence of hormonal effects on growth velocity and BMD; for children who may be entering puberty at or near upper end of this age bracket, puberty assessment will be based on clinical and laboratory findings 5. Must have received IV pamidronate therapy for at least one year prior to study initiation.

  * Type 3 OI will be confirmed with an Invitae Skeletal Dysplasia test, and clinical assessment including:

    * Blue/grey sclerae
    * Presence of prenatal fractures (on ultrasound when available)
    * Deformities present at birth (confirming prenatal fractures)
    * Severity of fractures and progressive deformities although no absolute 'number' of fractures is available

Exclusion Criteria:

1. Lacking confirmation of mutation in either COLA1A1 or COL1A2 genes
2. Other pathological types of OI
3. Any concurrent medical issue(s) known to decrease BMD (e.g., malabsorption conditions, glucocorticoid use)
4. Participation in other clinical trial
5. Vitamin D deficiency (<20 ng/dL) despite treatment
6. Clinically significant thrombocytopenia as defined by a platelet count of < 150,000x103/microliter ; anemia as defined by hemoglobin < 5th percentile for age (<11.5g/dL); neutropenia as defined by absolute neutrophil count < 1.5 x103/microliter; or elevations in the white blood cell count as defined by 3-6 year old-WBC > 15.5WBC x 103/microliter; 6-9 year old WBC >13.5 x103/microliter (Flerlage 2015)

8. PRA screening positive for anti-HLA antibodies 9. Elevated LFT's greater than 2 times the upper limit of normal 10. Other genetic disorders 11. Other skeletal dysplasia disorders 12. Other primary or secondary bone disorders 13. History of acute or chronic infections 14. History of cancer 15. History of thrombosis or prothrombotic disorders 16. History of heart disease 17. History of diabetes 18. History of strokes 19. History of vascular conditions 20. History of lung disease

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate of participants | Up to 24 months post-intervention
  Number of participants consented at the end of the trial
Number of participants with correctly collected data for the study outcomes | Up to 24 months post-intervention
  Number of participants with data correctly collected for the study outcomes
Total number of visits with protocol deviation | Up to 24 months post-intervention
  Total number of visits with protocol deviations at the end of the trial
Visit attendance by participants | Up to 1 year post last infusion intervention
  Percentage of visits completed by participants
Patient retention rate | Up to 1 year post last infusion intervention
  Percentage of patients that complete the study intervention and all follow up study visits
Patient Primary Clinical Outcome Retention Rate | Up to 1 year post last infusion intervention
  Percentage of participants that completed the primary clinical outcome measurements
Change in acceptability from baseline | Baseline, Up to 36 months post-intervention
  Acceptability will be evaluated with an end of study structured, verbal interview. This interview will consist of a mix of closed ended (scaled questions from 1[worst]-5 [best]) and open-ended questions giving subjective measurements. Open-ended questions will address overall experience during the study and prompt expression of thoughts or perspectives after completing the study. The total possible score range is 18 to 90. Higher score correlates with better outcome.
Number of unexpected adverse events | Up to 1 year post last infusion intervention
  Unexpected adverse events that occur from first study intervention to one year after last infusion.
Number of participants with change in vital signs from baseline | Baseline, 10 minutes pre-intervention, 15 minutes post-intervention, 30 minutes post-intervention, 1 hour post-intervention, 1 hour post completion of the infusion
  Number of participants with blood pressure, oxygen saturation, heart rate, respiratory rate, and temperature below or above each participants accepted mean reference range.
Number of participants with changes in laboratory panels from baseline (CBC, CMP) | Baseline, every 4 months post-intervention
  Number of patients with changes in CBC or CMP values from baseline CBC or CMP values. Any evidence of thrombocytopenia, anemia, neutropenia, or elevations in white blood counts will require consideration of stopping or pausing infusions by the PI. Slight changes in the ALT, AST, and calcium values are expected due to standard medication uses and will be monitored by PI.
Change in number of participants with changes in radiological parameters | Baseline, 8, 20 and 32 months post-intervention
  Number of participants with changes in radiological parameters (xrays and DXA scan) from baseline will be monitored during the study follow up time. DXA scans and x-rays used to assess for any semi-triggers that may require considerations of stopping or pausing infusions.
Change in annualized linear growth velocity | Baseline, every 4 months until 1 year after last infusion intervention
  This study will assess the annualized linear growth velocity at baseline and during cell therapy protocol in children with Type 3 OI (3-10 years of age and pre-pubertal at time of enrollment). Growth charts will be generated using growth measurements obtained every 4 months.
  Growth charts will be referenced against sex- and age-specific Centers for Disease Control and Prevention (CDC) childhood OI growth reference charts.
Change in fracture rate from baseline | Baseline, every 4 months post-intervention until 1 year after last infusion intervention
  Overt and covert fracture rate will be measured in each child at baseline and at regular intervals during MSC therapy by using a caretaker events diary, limb films, and spine films to tally more objectively new and healing fractures.
Change in bone mineral density from baseline | Baseline, yearly until 1 year after last infusion intervention
  Bone mineral density will be determined by DXA (dual-energy absorptiometry) analysis for TBLH (total body less head), spine and distal radius sites.
Change in bone age | Baseline, yearly until 1 year after last infusion intervention
  A bone age assessment is done using left hand radiograph. Bone age will be followed yearly in children of 8 years of age and older at time of enrollment in conjunction with exam and laboratory assessments to determine potential effects of puberty on bone density.
Change in Vertebral Compression Fractures (VCFs) | Baseline, every 18 months until one year after last infusion intervention
  Due to abnormal collagen and the associated decrease in BMD, VCFs are common in Type 3 OI. These can be 'silent' and/or associated with back pain. PA TL film and LAT TL film will be obtained to assess VCF's that cannot be assessed by DXA in children. Spine radiographs are within standard of care for treatment of OI.

SECONDARY OUTCOMES:
Number of participants with changes in bone metabolism markers | Baseline, every 12 months post-intervention, and at the conclusion of the study (up to 36 months post-intervention)
  Markers including osteocalcin, BAP, CTX, PICP, Calcium/Creatinine Ratio (urine), and NTX/Creatinine Ratio (urine) will be assessed for both bone health as well as bone formation/resorption.
Change in Limb Deformity Modified EOS Questionnaire (LD-EOSQ-22) from baseline | Baseline, annually until 1 year after last infusion
  This is a validated survey that will serve as a patient-reported outcome measure evaluating health status for these patients and the burden of their caregivers. The scores can range from 0-100 with a higher score correlating with a better outcome.
Change in BAMF (Brief Assessment of Motor Function) from baseline | Baseline, annually until 1 year after last infusion
  This validated survey contains 10 point ordinal scales that outline rapid descriptions for gross and fine motor performance. The higher you score on the BAMF survey, the more developed your gross and fine motor skills are.
Change in Pediatric Orthopedic Data Collection Instrument (PODCI) from baseline | Baseline, annually until 1 year after last intervention
  The PODCI questionnaire will used to quantify function abilities in our studied population. The scores can range from 0-100, with higher scores indicating higher levels of disability, and lower scores indicating better functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Doris Fadoju, MD, Principal Investigator — Emory University

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after de-identification and publication.
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following publication and then for a minimum of 5 years
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose, to achieve aims in the approved proposal.
  Proposals should be directed to edwin.horwitz@emory.edu. To gain access, data requestor will need to sign a data access agreement.